CLINICAL TRIAL: NCT05099692
Title: CHD Patient' s Concern on Primary Cardiac Rehabilitation and Its Social Associated Factors
Brief Title: CHD Patient's Concern on Cardiac Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Qiang Hu, Principal Investigator, Shenyang Northern Hospital
Other Study IDs: N2021-10
Record Dates: First submitted 2021-10-16; First posted 2021-10-29 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Coronary Heart Disease; Cardiac Rehabilitation
Keywords: cardiac rehabilitation; coronary heart disease; social-psychological factor
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHD patients participating in the cardiac rehabilitation
  Interventions: Behavioral: filling out the questionnaire

INTERVENTIONS:
Behavioral: filling out the questionnaire — all participants in our study are invited to choose at least 1 question in 15 questions or provide their own questions regarding their doubt about the CR after filling in their personal information

SUMMARY:
Our study focuses on the question about primary cardiac rehabilitation (CR) patients with coronary heart disease are concerned about demonstrating the association between the patients' view of CR and social associated factors. In our study, all participants are invited to choose at least 1 question in 15 questions or provide their questions regarding their doubt about the CR after filling in their personal information. The selectable questions can be categorized into five titles: the content or purpose of CR, the method of CR, the advantage of CR, the adverse effect of CR, and the expenditure of CR.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* patients diagnosed as coronary heart disease
* able to participate in cardiac rehabilitation after medical judgments for the first time
* understand the questionnaire content
* agree to participant in the study and provide the written informed consent

Exclusion Criteria:

* unable to complete the questionnaire
* patients who aren't willing or refuse to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease eligible for the study must be at least 18 years of age or greater, able to participate in cardiac rehabilitation after medical judgments by the physicians for the first time and provide the written informed consent. Moreover, the participants must understand the questionnaire content and complete it.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The total number of different selected questions | 5 minutes
  All participants are invited to choose at least 1 question in 15 questions or provide their questions regarding their doubt about the CR after filling in their personal information. As a result, we calculate and collect the total number of different selected questions for each patients.
The variety of different selected questions | 5 minutes
  All participants are invited to choose at least 1 question in 15 questions or provide their questions regarding their doubt about the CR after filling in their personal information. As a result, we calculate and collect the variety of different selected questions for each patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Qiang Hu, Shenyang, Liaoning, China